CLINICAL TRIAL: NCT00361855
Title: A Phase 1 Open Label Dose Escalation Study Evaluate The Safety Of a Single Escalating Dose Of NX-CP105 (Human Adult Bone Marrow Derived Somatic Cells [hABM-SC] Administered by Endomyocardial Injection To Cohorts Of Adults 30-60 Days Following Acute Myocardial Infarction
Brief Title: Safety Study of Bone Marrow Derived Cells to Treat Damaged Heart Muscle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuronyx (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-05-018
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Myocardial Infarction
Keywords: MI
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Drug: NX-CP105

SUMMARY:
Certain types of cells located in bone marrow may help the body recover after an injury. These cells may be able to help the body repair heart muscle that has been damaged from a heart attack. NX-CP105 is a new investigational drug that is made up of these special types of bone marrow cells, which come from another person. NX-CP105 has not been approved for sale or general use by the Food and Drug Administration (FDA), and this study will be the first time that NX-CP105 is given to human beings.

This study is being conducted to see if there are any side effects associated with with NX-CP105 and whether NX-CP105 may help the body repair heart muscle that has been damaged from a heart attack. Three different doses of NX CP105 will be tested in this study, starting with the lowest dose first.

Patients who decided to participate in the study will have a heart catheterization procedure during which a narrow tube is inserted into an artery (type of blood vessel) in the groin and passed to the heart. A second narrow tube will be inserted into a vein (type of blood vessel) in the groin and passed to your heart. A device will be passed through the second tube. This device will be used to inject NX-CP105 cells directly into your heart muscle.

DETAILED DESCRIPTION:
Each patient will go through three phases during the study. The first is the screening/baseline phase, the second is the treatment phase, and the third is the follow-up phase.

* The procedures that are required during the SCREENING/BASELINE PERIOD can be done in a doctor's office outside of the hospital.

  * Patients will be asked about their past medical conditions and the medicines you are taking.
  * Patients will be asked how often you get chest pain.
  * Patients will have a complete physical examination.
  * Patient vital signs (temperature, blood pressure, pulse and breathing rate) and weight will be measured.
  * Patients will give blood (about 2 tablespoons) and urine for routine laboratory tests, to see if you have been infected with certain viruses (HIV, Hepatitis B, Hepatitis C, CMV) and to test to determine blood type. A pregnancy test will be done if patients are capable of getting pregnant.
  * Patients will have an electrocardiogram (ECG - a painless heart beat tracing).
  * Patients will be asked to walk as fast as they can for six minutes.
  * Patients will have an x-ray type of test called a nuclear scan (SPECT) of your heart. A very small amount of a radioactive material will be injected into a vein during this test, which allows the doctor to evaluate blood flow in the heart.
  * Patients will have an echocardiogram, a procedure that uses sound waves to look at the position, size, and movement of heart valves and heart wall, as well as the direction of blood flow within the heart chambers. A solution that improves the ability of the echocardiogram device to look at the heart will be injected into a vein as part of this procedure.
  * Patients will be asked to wear a Holter monitor (a very small ECG machine) for 24 hours that will be worn around the neck in a Velcro pouch or in the shirt pocket. The monitor will be attached to the chest by three small adhesive patches and will be used to collect heart beat information. Patients will take off the patches after 24 hours and return the monitor to the study doctor.
* During the TREATMENT PERIOD patients will be kept in the hospital for at least 3 days during which they will receive the new investigational drug (NX-CP105).

  * Patients will need to be admitted to the hospital about a day before thet receive the study drug (bone marrow cells). During this time patients will have a procedure called cardiac catheterization. The study doctor will make a small puncture in the groin after the area is numbed with a local anesthetic (similar to Novocaine use by a dentist). Two thin catheters (tubes) will be placed in the groin area, one in a vein and one in an artery (large blood vessels). Blood thinners will be given during this procedure to help prevent blood clots. A series of thinner tubes (catheters) will then be inserted into the first tubes and will be carefully pushed up into the heart chambers. These catheters will be used to produce a 3-dimensional colored map (NOGA) that shows where the heart has been damaged. When mapping is complete, this catheter will be taken out and a new device with a needle in the tip will be run through the tubes. Using the map of your heart, the doctor will inject NX CP105 into parts of the heart that look like they were damaged.
  * After NX-CP105 is injected, all the tubes will be removed. After these procedures, patients will have another echocardiogram to look for heart or other problems that may have happened during the procedure. Patients will then be admitted to the intensive care unit (ICU) for at least 24 hours. Patients will remain in the hospital for at least 72 hours (3 days) after receiving NX-CP105.
  * Before leaving the hospital, patients will have another physical examination, including vital sign measurements and ECGs. Blood and urine laboratory safety samples will be collected
* The FOLLOW-UP PERIOD lasts 12 months. Patients will be asked to return to the study doctor for regular visits on Day 7, Day 14, Day 21, and 2 months, 3 months, 6 months and 12 months after receiving NX CP105. At each study visit, patients will be asked to do the following things:

  * Answer questions about any symptoms that you have had since the last study visit, including any chest pain.
  * Have a physical examination.
  * Have vital signs will be measured.
  * Give blood for routine laboratory tests.
  * Have an ECG.
  * Wear a Holter Monitor for 24 hours (except at the 6 and 12 month visits).
  * Have a six minute walk test (at the 3 and 6 month visits only).
  * Have a nuclear scan (SPECT) of the heart (at the 3 and 6 month visits only).
  * Have an echocardiogram (at the 3 and 6 month visits only).
  * Patients will also be admitted to the hospital to have another cardiac catheterization and NOGA mapping procedure when you come back for the 3 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* 30-75 years of age (inclusive)
* 30-60 days since AMI (defined as the most recent MI causing a doubling in cTnI enzyme concentrations relative to normal levels in addition to ECG changes consistent with MI with confirmation by myocardial perfusion imaging [SPECT])
* Successful percutaneous revascularization restoring TIMI II or higher flow to infarcted area
* Negative pregnancy test (serum βhCG) in women of childbearing potential (within 24 hours prior to dosing)
* LVEF ≥ 30% as measured by myocardial perfusion imaging (SPECT)
* Cardiac enzyme tests (CPK, CPK MB, cTnI) within the normal range at baseline
* Willing and able to comply with protocol, including follow-up visits
* Signed Subject Informed Consent Form

Exclusion Criteria:

* Significant coronary artery stenosis that may require percutaneous or surgical revascularization within six months of enrollment, as determined by the principal investigator
* LV thrombus (mobile or mural)
* High grade atrioventricular block (AVB)
* Frequent, recurrent, sustained (>30 seconds) or non-sustained ventricular tachycardia > 48 hours after AMI
* Clinically significant ECG abnormalities that may interfere with subject safety during the intracardiac mapping and injection procedure
* Atrial fibrillation with uncontrolled heart rate
* Severe valvular disease (e.g., aortic stenosis, mitral stenosis, severe valvular insufficiency requiring valve replacement)
* History of heart valve replacement
* Idiopathic cardiomyopathy
* Severe peripheral vascular disease
* Liver enzymes (aspartate aminotransferase [AST]/ alanine aminotransferase [ALT]) ≥ 3 times upper limit of normal (ULN)
* Serum creatinine ≥ 2.0 mg/dL
* History of active cancer within the preceding three years (with exception of basal cell carcinoma)
* Previous bone marrow transplant
* Known human immunodeficiency virus (HIV) infection
* Evidence of concurrent infection or sepsis on chest X-ray (CXR) or blood culture
* Participation in an experimental clinical trial within 30 days prior to enrollment
* Alcohol or recreational drug abuse within six months prior to enrollment
* Major surgical procedure or major trauma within the 14 days prior to enrollment
* Known autoimmune disease (e.g., systemic lupus erythematosus [SLE], multiple sclerosis)
* Clinically significant elevations in PT or PTT relative to laboratory norms
* Thrombocytopenia (platelet count < 50,000/mm3)
* Inadequately controlled diabetes mellitus type I or type II, defined as a change in anti-diabetic medication regimen within the prior 3 months or HbA1C > 7.0%
* Uncontrolled hypertension defined as systolic blood pressure (SBP) > 180 mmHg and/or diastolic blood pressure (DBP) >100 mmHg
* Use of ionotrophic drugs > 24 hours post AMI
* Other co-morbid conditions such as hemodynamic instability, unstable arrythmias, and intubation, which, in the opinion of the principal investigator, may place subjects at undue risk or interfere with the objectives of the study
* Any other major illness, which, in the opinion of the principal investigator, may interfere with the subject's ability to comply with the protocol, compromise subject safety, or interfere with the interpretation of the study results

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Safety as measured by clinical laboratory values, vital signs,
ECG/holter monitoring, echocardiogram

SECONDARY OUTCOMES:
Efficacy as measured by cardiac output/pressure gradients, myocardial perfusion, viability and ejection fraction,
BNP, six minute walk test, and remodeling by contrast enhance echocardiogram

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Heart Institute, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - Northwestern University, Chicago, Illinois
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania